CLINICAL TRIAL: NCT02566460
Title: The Effect of Lactate Clearance Oriented Haemodynamic Therapy on the Outcome of Patients With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PUMCH-S616
Record Dates: First submitted 2015-09-26; First posted 2015-10-02 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-02

CONDITIONS: Septic Shock
Keywords: Lactate clearance; systemic central venous oxygen saturation; septic shock; haemodynamic therapy
MeSH Terms: conditions — Shock, Septic | interventions — Resuscitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- lactate clearance group (Experimental): Refer to lactate clearance rate to perform resuscitation therapy
  Interventions: Other: Resuscitation
- SCVO2 group (Sham Comparator): Refer to SCVO2 to perform resuscitation therapy
  Interventions: Other: Resuscitation

INTERVENTIONS:
Other: Resuscitation — First, either crystalloid or colloid could be given to achieve a CVP of 8 to 12 mm Hg. Second, if the mean arterial pressure (MAP) was less than 65 mm Hg, norepinephrine was administrated to maintain MAP ≥65 mm Hg. If the mean arterial pressure was higher than 90 mm Hg, vasodilators were given until it was 90 mm Hg or below. Finally, SCVO2 or lactate clearance will be checked to determine red blood cells transfused or not to achieve a haematocrit of at least 30%. If ScvO2 or lactate clearance remains unmet target value, dobutamine could be used in the treatment.

SUMMARY:
The purpose of this study is to explore and assess possible outcome benefits of lactate clearance>30% vs ScvO2 ≥70% in 6 hours as the protocol goal that evaluated adequacy of during early resuscitation of septic shock through a single-center randomized controlled study. The investigators anticipate to collect 300-400 qualified patients with septic shock who were selected from critically ill patients admitted to the Department of Critical Care Medicine. The participants can be randomized divided into lactate clearance group and SCVO2 group. The investigators compared the treatment and the relevant parameters changed after different target. 28-day mortality, ICU and hospital lengths of stay, ventilator-free days, and new emerged organ failure were collected and compared. 28-day survival curves were drew between these two group. And the adverse events of the treatment have also been compared. Through this study, the investigators want to answer that whether lactate clearance-oriented therapy can reduce the mortality in patients with septic shock, compared with ScvO2-oriented protocolised therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with septic shock were assessed for inclusion, which required that patients be older than 18 years with confirmed or presumed infection, met two or more criteria for systemic inflammatory response syndrome [16], and evidence of refractory hypotension or a serum lactate level above 4 mmol per liter.
* Refractory hypotension was defined as a systolic blood pressure lower than 90 mm Hg, or a mean arterial pressure of less than 65 mm Hg , after an intravenous fluid challenge of 20 ml or more per kilogram of body weight.
* Patients had to be enrolled in the study within 2 hours after the earliest detection of septic shock and within 12 hours after arrival ICU.

Exclusion Criteria:

* The patients were excluded if they meet any one of follows: an age of less than 18 years, pregnancy, an acute cerebral vascular event (Glasgow coma score < 5), acute myocardial infarction or acute coronary syndrome, massive pulmonary embolism, status asthmaticus, a primary diagnosed cardiac dysrhythmias, contraindication to central venous catheterization, active gastrointestinal hemorrhage, massive intra abdominal infective focus without drainage, severe bronchopleural fistula, seizure, during chemotherapy or immunosuppressive therapy, or end stage of the diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
60-day mortality | 60 days

SECONDARY OUTCOMES:
ventilator-free days | 60 days
organs dysfunction/failure | 60 days
  New onset organs dysfunction/failure were defined with reference to internationally accepted criteria as follows. (1) In accordance with the RIFLE criteria, acute kidney injure (AKI) defined as the sudden changes (48 hours) of renal function caused by renal structural or function damaged, showing absolute increase in serum creatinine ≥0.3 mg / dl (≥26.4umol / l), or an increase ≥50% (1.5 times the baseline value), or urine output <0.5 ml/kg/h for over 6 hours. (2) Acute liver injury is defined as ALT increased more than 1 times. (3) Acute myocardial injury is defined as emerging symptoms of myocardial ischemia. ECG changes suggested myocardial ischemia (ST segment elevation or depression, or pathologic Q waves), and biochemical markers of myocardial necrosis was typical increased (troponin and creatine kinase). (4) Based on the Berlin definition, acute lung injury is defined as oxygenation index <300mmHg with PEEP ≥5 cmH2O.
the adverse events of the treatment | 60 days
  Acute pulmonary edema, Acute myocardial infarction, Arrhythmia, Cardiac Arrest, Pneumothorax caused by the puncture, RBC allergy, Catheter-related infections

REFERENCES:
- [Derived] Zhou X, Liu D, Su L, Yao B, Long Y, Wang X, Chai W, Cui N, Wang H, Rui X. Use of stepwise lactate kinetics-oriented hemodynamic therapy could improve the clinical outcomes of patients with sepsis-associated hyperlactatemia. Crit Care. 2017 Feb 16;21(1):33. doi: 10.1186/s13054-017-1617-1. PMID 28202033